CLINICAL TRIAL: NCT06511388
Title: Cardiotoxic Effects of Chemotherapy in Patients With Sarcomas: A Two and Three-Dimensional Echocardiographic Speckle Tracking Imaging Study
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 15-002714; NCI-2024-05323 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-002714 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-06-28; First posted 2024-07-22 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients receive anthracycline once a day or split between 2-3 days per SOC. Patients undergo 2D-STE throughout the study and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to identify markers that will allow researchers to identify in advance patients with sarcomas who are at highest risk for developing heart failure related to chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To detect acute and subacute changes in myocardial function by two-dimensional (2D)-Speckle Tracking Echocardiography (STE) derived strain and strain rate in sarcoma patients undergoing chemotherapeutic treatment.

Ia. To compare 2D-STE and three-dimensional (3D)-STE derived strain and strain-rate; Ib. To compare 2D-STE and 2D- and 3D-left ventricle ejection fraction (LVEF); Ic. If feasible, to compare 2D-STE and cardiac biomarkers [serum cardiac troponin T and N-terminal fragment of brain natriuretic peptide (NT-proBNP)].

II. To predict chemotherapy-induced cardiotoxicity by using 2D-STE and/or other significant parameters for early detection of cardiac dysfunction.

OUTLINE: This is an observational study.

Patients receive anthracycline once a day or split between 2-3 days per standard of care (SOC). Patients undergo 2D-STE throughout the study and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed at Mayo Clinic and treated for sarcoma with doxorubicin as first-line treatment

Exclusion Criteria:

* First-line treatment not including doxorubicin

  * Treatment performed outside of Mayo Clinic with different protocols
  * Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of sarcoma undergoing chemotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-01-20 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Changes in myocardial function - 2D-STE | Baseline, 3 months, 6 months, 1 year
  Changes in myocardial function will be assessed using 2D-STE derived strain rate. Changes will be compared to baseline over time.
Changes in myocardial function - 2D-STE vs 3D-STE | Baseline, 3 months, 6 months, 1 year
  Differences between two-dimensional speckle tracking echocardiography (2D-STE) and three-dimensional speckle tracking echocardiography (3D-STE) derived strain will be compared at baseline and over time.
Changes in myocardial function - 2D-STE vs 2D-LVEF and 3D-LVEF | Baseline, 3 months, 6 months, 1 year
  Differences between 2D-STE and 2D- and 3D- left ventricle ejection fraction (2D-LVEF and 3D-LVEF, respectively) will be compared at baseline and over time.
Changes in myocardial function - 2D-STE vs cardiac biomarkers | Baseline, 3 months, 6 months, 1 year
  If feasible, 2D-STE and cardiac biomarkers [serum cardiac troponin T and N-terminal fragment of brain natriuretic peptide (NT-proBNP)] will be compared at baseline and over time.

CONTACTS AND LOCATIONS:
Overall Officials: Hector R. Villarraga, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials